CLINICAL TRIAL: NCT02949726
Title: Lymphatic and Systemic Immunity Changes in Post-radiation Lymphedema Development
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: M.D. Anderson Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa B Aldrich, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-15-1021; 1R01CA201487-01A1 (NIH)
Record Dates: First submitted 2016-07-11; First posted 2016-10-31 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Cancer-treated patients receiving NIRFLI (Other): Near-infrared Fluorescence Lymphatic Imaging (NIRFLI) using Indocyanine Green (ICG) is used to "visualize" lymphatic vessel anatomy and function.
  Interventions: Drug: Indocyanine Green (ICG); Device: Near-infrared Fluorescence Lymphatic Imaging (NIRFLI)

INTERVENTIONS:
Drug: Indocyanine Green (ICG) — Near-infrared Fluorescence Lymphatic Imaging (NIRFLI) using Indocyanine Green (ICG) is used to "visualize" lymphatic vessel anatomy and function.
Device: Near-infrared Fluorescence Lymphatic Imaging (NIRFLI) — Near-infrared Fluorescence Lymphatic Imaging (NIRFLI) using Indocyanine Green (ICG) is used to "visualize" lymphatic vessel anatomy and function.

SUMMARY:
The goal of this study is to find out which immune molecules, cells, and genes are involved in the development of lymphedema (LE), so that medicines that target them can be considered for treating lymphedema. The hypothesis is that LE is a systemic, autoimmune-like disease that is initiated by inflammatory cytokines induced by surgery, radiation, and possibly chemotherapy in genetically susceptible patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* Participants must have been clinically diagnosed with breast cancer and scheduled for axillary lymph node dissection (ALND) and radiation treatment at MD Anderson (receiving chemotherapy, mastectomy or breast-conserving surgery, ALND (>10 nodes) and radiation treatment for breast cancer, identified by Drs. Mittendorf and Shaitelman of the Nellie B. Connally Breast Cancer Center at MD Anderson)
* Ambulatory and possessing all four limbs
* No prior radiation therapy
* Negative urine pregnancy test within 36 hours prior to study drug administration, if of childbearing potential
* Females participants must complete the Female Enrollment Form. Childbearing potential participants must agree to use one of the medically accepted forms of contraception for a period of one month after study participation. Female participants who meet the criteria for non-childbearing will still complete the Female Enrollment Form, but are not restricted to the use of contraception following study participation.

Exclusion Criteria:

* Participants with a known or suspected allergy to iodine
* Participants who are breastfeeding, pregnant or trying to become pregnant
* Severe underlying chronic illness or disease (other than breast cancer)
* Participants not capable of keeping moderately still for the imaging portion of the study session (~1 hour for imaging)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Lymphatic propulsive velocity as assessed by NIRFLI | immediately before surgery
Lymphatic propulsive velocity as assessed by NIRFLI | immediately before radiation (which is 6-8 weeks after surgery)
Lymphatic propulsive velocity as assessed by NIRFLI | 6 months after radiation
Lymphatic propulsive velocity as assessed by NIRFLI | 12 months after radiation
Lymphatic propulsive velocity as assessed by NIRFLI | 24 months after radiation
Lymphatic propulsive frequency as assessed by NIRFLI | immediately before surgery
Lymphatic propulsive frequency as assessed by NIRFLI | immediately before radiation (which is 6-8 weeks after surgery)
Lymphatic propulsive frequency as assessed by NIRFLI | 6 months after radiation
Lymphatic propulsive frequency as assessed by NIRFLI | 12 months after radiation
Lymphatic propulsive frequency as assessed by NIRFLI | 24 months after radiation
Percent extravascular dye as assessed by NIRFLI | immediately before surgery
Percent extravascular dye as assessed by NIRFLI | immediately before radiation (which is 6-8 weeks after surgery)
Percent extravascular dye as assessed by NIRFLI | 6 months after radiation
Percent extravascular dye as assessed by NIRFLI | 12 months after radiation
Percent extravascular dye as assessed by NIRFLI | 24 months after radiation
Vessel tortuosity as assessed by NIRFLI | immediately before surgery
Vessel tortuosity as assessed by NIRFLI | immediately before radiation (which is 6-8 weeks after surgery)
Vessel tortuosity as assessed by NIRFLI | 6 months after radiation
Vessel tortuosity as assessed by NIRFLI | 12 months after radiation
Vessel tortuosity as assessed by NIRFLI | 24 months after radiation
Vessel dilation ratio as assessed by NIRFLI | immediately before surgery
Vessel dilation ratio as assessed by NIRFLI | immediately before radiation (which is 6-8 weeks after surgery)
Vessel dilation ratio as assessed by NIRFLI | 6 months after radiation
Vessel dilation ratio as assessed by NIRFLI | 12 months after radiation
Vessel dilation ratio as assessed by NIRFLI | 24 months after radiation

SECONDARY OUTCOMES:
Chemokine levels as assessed by bead assay | immediately before surgery
Chemokine levels as assessed by bead assay | immediately before radiation (which is 6-8 weeks after surgery)
Chemokine levels as assessed by bead assay | 6 months after radiation
Chemokine levels as assessed by bead assay | 12 months after radiation
Chemokine levels as assessed by bead assay | 24 months after radiation
Cytokine levels as assessed by bead assay | immediately before surgery
Cytokine levels as assessed by bead assay | immediately before radiation (which is 6-8 weeks after surgery)
Cytokine levels as assessed by bead assay | 6 months after radiation
Cytokine levels as assessed by bead assay | 12 months after radiation
Cytokine levels as assessed by bead assay | 24 months after radiation
Number of participants with autoimmune antibodies as assessed by ELISA | immediately before surgery
Number of participants with autoimmune antibodies as assessed by ELISA | immediately before radiation (which is 6-8 weeks after surgery)
Number of participants with autoimmune antibodies as assessed by ELISA | 6 months after radiation
Number of participants with autoimmune antibodies as assessed by ELISA | 12 months after radiation
Number of participants with autoimmune antibodies as assessed by ELISA | 24 months after radiation

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Aldrich, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States